CLINICAL TRIAL: NCT05742477
Title: Treatment Outcome With Antibiotic Use and Its Resistance Pattern Among Patient With Neonatal Sepsis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abd elrahman Ahmed Hussain Abd eltwaab, Principal investigator, Assiut University
Other Study IDs: neonatal sepsis treatment
Record Dates: First submitted 2022-08-22; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Neonatal Sepsis
Keywords: neonatal; sepsis; antibiotics
MeSH Terms: conditions — Neonatal Sepsis; Sepsis | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antibiotic — role of antibiotics in treatment of neonatal sepsis

SUMMARY:
Determine Treatment outcome with antibiotic use and its resistance pattern among neonatal sepsis patients

DETAILED DESCRIPTION:
Neonatal sepsis is a clinical syndrome characterized by systemic signs and symptoms of infection and is accompanied by bacteremia in the first month of life. Early-onset sepsis (EOS) is defined as sepsis occurring in the first 72 h of life and that occurring beyond 72 h is defined as late-onset sepsis (LOS). As per World Health Organization (WHO), neonatal sepsis is the third most frequent etiology of neonatal mortality. In the year 2013, a systematic analysis of global, national, and regional causes of child mortality found neonatal sepsis to be the leading cause of neonatal deaths in Europe. The National Neonatal Perinatal Database network (NNPD, 2002-03) comprising 18 tertiary care neonatal units across Europe reported sepsis (septicemia/meningitis) as the commonest cause of neonatal mortality, causing 23.4% of all neonatal deaths. The pattern of the bacterial pathogens responsible for neonatal sepsis has changed temporally and geographically. There is a difference in the causative organisms for neonatal sepsis between developed and developing countries. As per NNPD, Klebsiella pneumonia and Staphylococcus aureus are the commonest causative organisms for EOS and LOS in Europe. On the contrary, data from developed countries shows that gram-positive organisms are the predominant causes of EOS as well as LOS. The ability of bacteria to resist or to become tolerant to several structurally and functionally distinct drugs simultaneously is known as multidrug resistance. Simpler definitions quote "multidrug-resistant organisms (MDROs) are labeled as such because of their in-vitro resistance to more than one antimicrobial agent". On the other hand, definitions vary per specific organism. It is estimated that in Europe, 56,524 neonatal deaths each year are attributed to isolates resistant to first-line antibiotics. A recent point prevalence study - Antibiotic Resistance and Prescribing in European Children (ARPEC) was conducted in 226 hospitals (41 countries) which. This survey showed that most commonly used regimen for neonatal sepsis was a combination of ampicillin/amoxicillin/benzylpenicillin Faculty of Medicine Institutional Review Board (IRB) Assiut Medical School Research Proposal Form 3 and aminoglycoside. It further reported that 40% of pathogens isolated were resistant to first-line antibiotics prescribed by WHO. Though this survey had a paucity of data from low- and middle-income countries (LMICs), it provided important insights into the emergence of antibiotic resistance. Resistance to first-line antibiotics in different WHO regions Estimates of MDRO burden have also been reported from other countries. In a systematic review of five countries in South Asia (India, Pakistan, Sri Lanka, Bangladesh, and Nepal) comprising 109 studies, a high proportion of MDRO was reported. The pooled estimated data from hospitals and communities showed that Klebsiella pneumonia, E. coli, and Acinetobacter baumannii were multidrug resistant in 70.7%, 54%, and 78.7% of isolates respectively. A retrospective single-center study from Jordan evaluated 4 y data of 68 episodes of culture-positive neonatal sepsis. Gram-negative organisms were the commonest and 69% of these were multidrug resistant. In another cohort study from Taiwan, conducted over 8 y, 1106 episodes of culture-positive sepsis were reported. Of these, one-third were caused by gram-negative bacilli and 70 (18.6%) were multidrug resistant. A meta-analysis of 71 studies reported from China showed that 50% of gram-negative organisms were resistant to third-generation cephalosporins. Early signs of neonatal sepsis are : Diminished spontaneous activity Less vigorous sucking Anorexia Apnea Bradycardia Temperature instability (hypothermia or hyperthermia) Fever is present in only 10 to 15% of neonates but, when sustained (eg, > 1 hour), generally indicates infection. Other symptoms and signs include respiratory distress, neurologic findings (eg, seizures,itteriness), jaundice (especially occurring within the first 24 hours of life without Rh or ABO blood group incompatibility and with a higher than expected direct bilirubin concentration), vomiting, diarrhea, and abdominal distention. Periumbilical erythema, discharge, or bleeding without a hemorrhagic diathesis suggests omphalitis Faculty of Medicine Institutional Review Board (IRB) Assiut Medical School Research Proposal Form 4 (infection prevents obliteration of the umbilical vessels). Coma, seizures, opisthotonos, or a bulging fontanelle suggests meningitis, encephalitis, or brain abscess.

Decreased spontaneous movement of an extremity and swelling, warmth, erythema, or tenderness over a joint indicates osteomyelitis or pyogenic arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Newborn suspected with sepsis diagnosed on the basis of clinical signs and symptoms:
* temperature instability
* feeding problems,
* convulsions,
* lethargy
* respiratory distress.
* laboratory findings such as:
* C-Reactive Protein (CRP)
* complete blood count (CBC)
* blood/urine cultures

Exclusion Criteria:

* Respiratory distress syndrome
* Congenital pneumonia

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients with neonatal sepsis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-31 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Sepsis convelence | 24hours
  It is difined by abcence of fever, jundice, respiratory failure and gastroentritis
Sepsis convelence | 1 week
  It is difined by abcence of fever, jundice, respiratory failure and gastroentritis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klein JO. Bacteriology of neonatal sepsis. Pediatr Infect Dis J. 1990 Oct;9(10):778. No abstract available. PMID 2235163
- [Background] Liu L, Oza S, Hogan D, Chu Y, Perin J, Zhu J, Lawn JE, Cousens S, Mathers C, Black RE. Global, regional, and national causes of under-5 mortality in 2000-15: an updated systematic analysis with implications for the Sustainable Development Goals. Lancet. 2016 Dec 17;388(10063):3027-3035. doi: 10.1016/S0140-6736(16)31593-8. Epub 2016 Nov 11. PMID 27839855
- [Background] Liu L, Johnson HL, Cousens S, Perin J, Scott S, Lawn JE, Rudan I, Campbell H, Cibulskis R, Li M, Mathers C, Black RE; Child Health Epidemiology Reference Group of WHO and UNICEF. Global, regional, and national causes of child mortality: an updated systematic analysis for 2010 with time trends since 2000. Lancet. 2012 Jun 9;379(9832):2151-61. doi: 10.1016/S0140-6736(12)60560-1. Epub 2012 May 11. PMID 22579125
- [Background] Stoll BJ, Hansen NI, Sanchez PJ, Faix RG, Poindexter BB, Van Meurs KP, Bizzarro MJ, Goldberg RN, Frantz ID 3rd, Hale EC, Shankaran S, Kennedy K, Carlo WA, Watterberg KL, Bell EF, Walsh MC, Schibler K, Laptook AR, Shane AL, Schrag SJ, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Early onset neonatal sepsis: the burden of group B Streptococcal and E. coli disease continues. Pediatrics. 2011 May;127(5):817-26. doi: 10.1542/peds.2010-2217. Epub 2011 Apr 25. PMID 21518717
- See also: Early onset neonatal sepsis: the burden of group B Streptococcal and E. coli disease continues — https://pubmed.ncbi.nlm.nih.gov/21518717/